CLINICAL TRIAL: NCT01252355
Title: A Multi-center Double-blind Parallel-group Placebo-controlled Study of the Efficacy and Safety of Teriflunomide in Patients With Relapsing Multiple Sclerosis Who Are Treated With Interferon-beta
Brief Title: Efficacy and Safety of Teriflunomide in Patients With Relapsing Multiple Sclerosis and Treated With Interferon-beta
Acronym: TERACLES
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision to prematurely stop the study, not linked to any safety concern.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC6058; 2010-023172-12 (EudraCT Number); U1111-1115-2414 (Other: UTN)
Record Dates: First submitted 2010-11-30; First posted 2010-12-03 (Estimated); Results first posted 2014-05-22 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Multiple Sclerosis Relapse
MeSH Terms: interventions — teriflunomide; Interferon-beta

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Teriflunomide 7 mg + IFN-beta (Experimental): Teriflunomide 7 milligram (mg) once a day concomitantly with IFN-beta therapy.
  Interventions: Drug: Teriflunomide; Drug: Interferon-beta (IFN-beta)
- Teriflunomide 14 mg + IFN-beta (Experimental): Teriflunomide 14 mg once a day concomitantly with IFN-beta therapy.
  Interventions: Drug: Teriflunomide; Drug: Interferon-beta (IFN-beta)
- Placebo + IFN-beta (Placebo Comparator): Placebo (for teriflunomide) once a day concomitantly with IFN-beta therapy.
  Interventions: Drug: Placebo (for teriflunomide); Drug: Interferon-beta (IFN-beta)

INTERVENTIONS:
Drug: Teriflunomide — Film-coated tablet
  Oral administration
  Other Names: HMR1726
  Arms: Teriflunomide 14 mg + IFN-beta; Teriflunomide 7 mg + IFN-beta
Drug: Placebo (for teriflunomide) — Film-coated tablet
  Oral administration
  Arms: Placebo + IFN-beta
Drug: Interferon-beta (IFN-beta) — Any of the IFN-beta which are approved for marketed use in the country where the patient is enrolled.
  Administration according to the package insert.

SUMMARY:
The primary objective was to demonstrate the effect of teriflunomide, in comparison to placebo, on frequency of Multiple Sclerosis (MS) relapses in patients with relapsing forms of MS who are treated with Interferon-beta (IFN-beta).

The secondary objectives were:

* Assess the effect of teriflunomide, in comparison to placebo, when added to IFN-beta on:

  * Disease activity as measured by brain Magnetic Resonance Imaging (MRI)
  * Disability progression
  * Burden of disease and disease progression as measured by brain MRI
* Evaluate the safety and tolerability of teriflunomide when added to IFN-beta therapy
* Assess the pharmacokinetics of teriflunomide in use in addition to baseline IFN-beta therapy
* Assess associations between variations in genes and clinical outcomes (safety and efficacy)
* Assess other measures of efficacy of teriflunomide such as fatigue and health-related quality of life
* Assess measures of health economics (hospitalization due to relapse, including the length of stay and any admission to intensive care unit)

DETAILED DESCRIPTION:
The study period per patient was expected to be between 56 and 160 weeks depending on when the patient was randomized and this included the following:

* a screening period up to 4 weeks,
* a treatment period expected to be between 48 and 152 weeks,
* 4-week post rapid elimination follow-up period.

Patients were to continue on treatment until a fixed common end date which was approximately 48 weeks after randomization of the last patient.

For those patients who completed the treatment period, a long term extension study of approximately 1 year (including teriflunomide alone) was initially planned to be proposed.

ELIGIBILITY:
Inclusion criteria :

* Patient with relapsing forms of MS treated with IFN-beta
* Stable dose of IFN-beta (approved brand) for at least 6 months prior to randomization
* Disease activity in the 12 months prior to randomization and after first 3 months of IFN-beta treatment (defined by at least 1 relapse supported by EDSS or equivalent neurological examination, or, at least 1 brain or spinal cord MRI with at least one T1 gadolinium enhancing lesion)

Exclusion criteria:

* McDonald criteria for MS diagnosis not met at time of screening visit
* EDSS score greater than (>) 5.5 at randomization visit
* A relapse within 30 days prior randomization
* Persistent significant or severe infection
* Patients must not have used adrenocorticotrophic hormone or systemic corticosteroids for 2 weeks prior to randomization
* Prior or concomitant use of cytokine therapy (except baseline interferons), glatiramer acetate or intravenous immunoglobulins in the 3 months preceding randomization
* Liver function impairment or persisting elevations (confirmed by retest) of alanine aminotransferase (ALT), aspartate aminotransferase (AST), or direct bilirubin greater than 2 times the upper limit of normal range (ULN)
* Active hepatitis or hepatobiliary disease or known history of severe hepatitis
* Pregnant or breast-feeding women or those who were planning to become pregnant during the study
* Significantly impaired bone marrow function or significant anemia, leukopenia, or thrombocytopenia
* Human Immunodeficiency Virus (HIV) positive
* Known history of active tuberculosis not adequately treated
* Prior use within 2 years preceding randomization or concomitant use of cladribine and mitoxantrone
* Prior use within 6 months preceding randomization or concomitant use of natalizumab, or any other immunosuppressive agents such as azathioprine, cyclophosphamide, cyclosporine, methotrexate, mycophenolate, or fingolimod

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 534 (Actual)
Dates: Start 2011-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (185):
- United States (32):
  - Investigational Site Number 840049, Cullman, Alabama
  - Investigational Site Number 840005, Cordova, Alaska
  - Investigational Site Number 840003, Phoenix, Arizona
  - Investigational Site Number 840011, Oceanside, California
  - Investigational Site Number 840036, Fort Collins, Colorado
  - Investigational Site Number 840012, Maitland, Florida
  - Investigational Site Number 840013, Ormond Beach, Florida
  - Investigational Site Number 840055, Pompano Beach, Florida
  - Investigational Site Number 840021, St. Petersburg, Florida
  - Investigational Site Number 840004, Tampa, Florida
  - Investigational Site Number 840047, Tampa, Florida
  - Investigational Site Number 840034, Chicago, Illinois
  - Investigational Site Number 840037, Elk Grove Village, Illinois
  - Investigational Site Number 840033, Louisville, Kentucky
  - Investigational Site Number 840041, Baltimore, Maryland
  - Investigational Site Number 840028, Baltimore, Maryland
  - Investigational Site Number 840016, Clinton Township, Michigan
  - Investigational Site Number 840031, St Louis, Missouri
  - Investigational Site Number 840030, St Louis, Missouri
  - Investigational Site Number 840009, Missoula, Montana
  - Investigational Site Number 840023, Albuquerque, New Mexico
  - Investigational Site Number 840015, New York, New York
  - Investigational Site Number 840027, Charlotte, North Carolina
  - Investigational Site Number 840006, Bismarck, North Dakota
  - Investigational Site Number 840007, Fargo, North Dakota
  - Investigational Site Number 840046, Dayton, Ohio
  - Investigational Site Number 840017, Toledo, Ohio
  - Investigational Site Number 840043, Tulsa, Oklahoma
  - Investigational Site Number 840002, Nashville, Tennessee
  - Investigational Site Number 840040, Round Rock, Texas
  - Investigational Site Number 840020, San Antonio, Texas
  - Investigational Site Number 840032, Vienna, Virginia
- Argentina (3):
  - Investigational Site Number 032002, Argentina
  - Investigational Site Number 032003, Buenos Aires
  - Investigational Site Number 032004, Caba
- Australia (5):
  - Investigational Site Number 036008, Bedford Park
  - Investigational Site Number 036005, Chatswood
  - Investigational Site Number 036001, Heidelberg West
  - Investigational Site Number 036004, Kogarah
  - Investigational Site Number 036010, New Lambton
- Austria (2):
  - Investigational Site Number 040001, Graz
  - Investigational Site Number 040004, Linz
- Belgium (7):
  - Investigational Site Number 056005, Charleroi
  - Investigational Site Number 056004, Ghent
  - Investigational Site Number 056003, Hasselt
  - Investigational Site Number 056006, La Louvière
  - Investigational Site Number 056002, Leuven
  - Investigational Site Number 056001, Sijsele-Damme
  - Investigational Site Number 056007, Wilrijk
- Brazil (5):
  - Investigational Site Number 076009, Joinville
  - Investigational Site Number 076012, Passo Fundo
  - Investigational Site Number 076003, Porto Alegre
  - Investigational Site Number 076007, São Paulo
  - Investigational Site Number 076013, São Paulo
- Canada (9):
  - Investigational Site Number 124005, Calgary
  - Investigational Site Number 124004, Edmonton
  - Investigational Site Number 124003, Gatineau
  - Investigational Site Number 124006, Kingston
  - Investigational Site Number 124007, Montreal
  - Investigational Site Number 124008, Ottawa
  - Investigational Site Number 124002, Regina
  - Investigational Site Number 124001, Sherbrooke
  - Investigational Site Number 124009, Winnipeg
- Chile (3):
  - Investigational Site Number 152003, Santiago
  - Investigational Site Number 152004, Santiago
  - Investigational Site Number 152005, Viña del Mar
- Colombia (4):
  - Investigational Site Number 170001, Barranquilla
  - Investigational Site Number 170005, Bogotá
  - Investigational Site Number 170007, Bogotá
  - Investigational Site Number 170009, Medellín
- Investigational Site Number 208002, Aarhus C, Denmark
- Estonia (2):
  - Investigational Site Number 233002, Tallinn
  - Investigational Site Number 233001, Tartu
- Finland (5):
  - Investigational Site Number 246003, Helsinki
  - Investigational Site Number 246006, Hyvinkää
  - Investigational Site Number 246004, Oulu
  - Investigational Site Number 246002, Pori
  - Investigational Site Number 246001, Turku
- France (6):
  - Investigational Site Number 250003, Besançon
  - Investigational Site Number 250010, Clermont-Ferrand
  - Investigational Site Number 250002, Lyon
  - Investigational Site Number 250004, Montpellier
  - Investigational Site Number 250001, Nancy
  - Investigational Site Number 250006, Nantes
- Germany (23):
  - Investigational Site Number 276009, Bad Mergentheim
  - Investigational Site Number 276020, Bamberg
  - Investigational Site Number 276003, Bayreuth
  - Investigational Site Number 276015, Berlin
  - Investigational Site Number 276016, Berlin
  - Investigational Site Number 276021, Berlin
  - Investigational Site Number 276012, Bonn
  - Investigational Site Number 276005, Dresden
  - Investigational Site Number 276032, Düsseldorf
  - Investigational Site Number 276018, Erbach im Odenwald
  - Investigational Site Number 276004, Erlangen
  - Investigational Site Number 276028, Freiburg im Breisgau
  - Investigational Site Number 276006, Giessen
  - Investigational Site Number 276010, Hamburg
  - Investigational Site Number 276022, Hennigsdorf
  - Investigational Site Number 276024, Kassel
  - Investigational Site Number 276001, Leipzig
  - Investigational Site Number 276013, Mainz
  - Investigational Site Number 276023, Minden
  - Investigational Site Number 276002, Münster
  - Investigational Site Number 276031, Rostock
  - Investigational Site Number 276008, Wiesbaden
  - Investigational Site Number 276026, Wuppertal
- Greece (4):
  - Investigational Site Number 300002, Athens
  - Investigational Site Number 300001, Athens
  - Investigational Site Number 300003, Heraklion
  - Investigational Site Number 300006, Thessaloniki
- Hungary (8):
  - Investigational Site Number 348002, Budapest
  - Investigational Site Number 348006, Budapest
  - Investigational Site Number 348010, Budapest
  - Investigational Site Number 348009, Eger
  - Investigational Site Number 348003, Esztergom
  - Investigational Site Number 348001, Szeged
  - Investigational Site Number 348005, Székesfehérvár
  - Investigational Site Number 348007, Zalaegerszeg
- Italy (11):
  - Investigational Site Number 380009, Catania
  - Investigational Site Number 380002, Cefalù
  - Investigational Site Number 380003, Fidenza
  - Investigational Site Number 380004, Gallarate
  - Investigational Site Number 380012, Montichiari
  - Investigational Site Number 380010, Napoli
  - Investigational Site Number 380011, Napoli
  - Investigational Site Number 380006, Padua
  - Investigational Site Number 380005, Roma
  - Investigational Site Number 380008, Roma
  - Investigational Site Number 380014, Verona
- Lithuania (3):
  - Investigational Site Number 440002, Kaunas
  - Investigational Site Number 440004, Klaipėda
  - Investigational Site Number 440003, Šiauliai
- Netherlands (4):
  - Investigational Site Number 528001, Breda
  - Investigational Site Number 528005, Nieuwegein
  - Investigational Site Number 528002, Sittard-Geleen
  - Investigational Site Number 528006, Venray
- Investigational Site Number 578002, Tønsberg, Norway
- Portugal (4):
  - Investigational Site Number 620001, Amadora
  - Investigational Site Number 620002, Coimbra
  - Investigational Site Number 620004, Coimbra
  - Investigational Site Number 620003, Setúbal
- Russia (17):
  - Investigational Site Number 643012, Kaluga
  - Investigational Site Number 643007, Kazan'
  - Investigational Site Number 643001, Kemerovo
  - Investigational Site Number 643013, Moscow
  - Investigational Site Number 643006, Nizhny Novgorod
  - Investigational Site Number 643004, Nizhny Novgorod
  - Investigational Site Number 643015, Novosibirsk
  - Investigational Site Number 643010, Rostov-on-Don
  - Investigational Site Number 643009, Rostov-on-Don
  - Investigational Site Number 643011, Saint Petersburg
  - Investigational Site Number 643018, Saint Petersburg
  - Investigational Site Number 643003, Saint Petersburg
  - Investigational Site Number 643017, Saint Petersburg
  - Investigational Site Number 643002, Saint Petersburg
  - Investigational Site Number 643016, Samara
  - Investigational Site Number 643005, Smolensk
  - Investigational Site Number 643014, Yaroslavl
- Slovakia (2):
  - Investigational Site Number 703002, Martin
  - Investigational Site Number 703001, Trnava
- South Korea (3):
  - Investigational Site Number 410002, Goyang-si
  - Investigational Site Number 410004, Seoul
  - Investigational Site Number 410001, Seoul
- Spain (8):
  - Investigational Site Number 724001, Barcelona
  - Investigational Site Number 724002, Barcelona
  - Investigational Site Number 724009, Córdoba
  - Investigational Site Number 724003, Girona
  - Investigational Site Number 724004, Madrid
  - Investigational Site Number 724005, Madrid
  - Investigational Site Number 724007, Murcia
  - Investigational Site Number 724008, Seville
- Sweden (3):
  - Investigational Site Number 752004, Gothenburg
  - Investigational Site Number 752003, Stockholm
  - Investigational Site Number 752001, Stockholm
- Tunisia (4):
  - Investigational Site Number 788002, Manouba
  - Investigational Site Number 788005, Monastir
  - Investigational Site Number 788004, Sfax
  - Investigational Site Number 788006, Tunis
- United Kingdom (6):
  - Investigational Site Number 826008, Birmingham
  - Investigational Site Number 826005, Leeds
  - Investigational Site Number 826006, Liverpool
  - Investigational Site Number 826003, London
  - Investigational Site Number 826004, Plymouth
  - Investigational Site Number 826001, Salford

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment initiated in January 2011, was discontinued in December 2012 following the decision of the Sponsor to discontinue the study, the common treatment end date was defined as February 28th, 2013 (treatment duration between 24 and 108 weeks).
  A total of 846 participants were screened at 185 sites in 28 countries.
Pre-assignment Details: Randomization was stratified by investigational site and Interferon-beta (IFN-beta) dose level (high/low). Assignment to groups was done centrally using an Interactive Voice Response System (IVRS) in a 1:1:1 ratio after confirmation of selection criteria. A total of 534 participants were randomized.
Groups:
- Placebo + IFN-beta: Placebo (for teriflunomide) once daily concomitantly with IFN-beta.
- Teriflunomide 7 mg + IFN-beta: Teriflunomide 7 mg once daily concomitantly with IFN-beta.
- Teriflunomide 14 mg + IFN-beta: Teriflunomide 14 mg once daily concomitantly with IFN-beta.
Period: Overall Study
Arm/Group | Placebo + IFN-beta | Teriflunomide 7 mg + IFN-beta | Teriflunomide 14 mg + IFN-beta
Started | 177 (Randomized.) | 178 (Randomized.) | 179 (Randomized.)
Treated | 175 | 178 | 179 (One participant received teriflunomide 7 mg.)
Completed | 0 | 0 | 0
Not Completed | 177 | 178 | 179
Not completed — Adverse Event | 9 | 17 | 22
Not completed — Lack of Efficacy | 6 | 4 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Poor Compliance to Protocol | 1 | 1 | 1
Not completed — Progressive Disease | 2 | 0 | 0
Not completed — Sponsor Early Termination of Study | 149 | 149 | 146
Not completed — Randomized but not Treated | 2 | 0 | 0
Not completed — Other Than Above | 8 | 7 | 7

BASELINE CHARACTERISTICS:
Population: Randomized population: all randomized participants according to the treatment group to which they were assigned.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + IFN-beta | Teriflunomide 7 mg + IFN-beta | Teriflunomide 14 mg + IFN-beta | Total
Number analyzed (Participants) | 177 | 178 | 179 | 534
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (8.9) | 38.7 (9.5) | 37.7 (9.2) | 38.2 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 125 | 114 | 352
  Male | 64 | 53 | 65 | 182
Region of Enrollment [Number; unit: participants] — Due to the small sample size in some countries, the countries were pooled as follows:
  * America: Argentina, Brazil, Canada, Chile, Columbia, The United States
  * Western Europe: Austria, Belgium, Denmark, Finland, France, Germany, Italy, Netherlands, Norway, Portugal, Spain, Sweden, The United Kingdom
  * Eastern Europe = Estonia, Greece, Hungary, Lithuania, Russian Federation, Slovakia
  * Asia, Africa and Australia = Australia, Republic of Korea, Tunisia
  participants
    America | 33 | 30 | 37 | 100
    Western Europe | 86 | 86 | 79 | 251
    Eastern Europe | 51 | 51 | 56 | 158
    Asia, Africa and Australia | 7 | 11 | 7 | 25
Time Since First Diagnosis of Multiple Sclerosis (MS) [Mean (Standard Deviation); unit: years] | 7.0 (5.6) | 6.6 (5.6) | 6.8 (5.9) | 6.8 (5.7)
Number of MS Relapses [Median (Full Range); unit: MS relapses] — The information was not available for one participant in the "Teriflunomide 14 mg + IFN-beta" group.
  MS relapses
    Within the past year | 1 [0 to 4] | 1 [0 to 3] | 1 [0 to 4] | 1 [0 to 4]
    Within the past 2 years | 2 [0 to 6] | 2 [0 to 8] | 2 [0 to 8] | 2 [0 to 8]
Time Since Most Recent MS Relapse Onset [Median (Full Range); unit: months] | 5.0 (8.29) [1.0 to 75.0] | 5.0 (4.83) [1.0 to 36.0] | 4.0 (15.36) [1.0 to 174.0] | 5.0 (10.47) [1.0 to 174.0]
MS Subtype [Number; unit: participants]
  Relapsing Remitting | 174 | 173 | 175 | 522
  Secondary Progressive | 2 | 3 | 4 | 9
  Progressive Relapsing | 1 | 2 | 0 | 3
Baseline Expanded Disability Status Scale (EDSS) Score [Mean (Standard Deviation); unit: units on a scale] — EDSS is an ordinal scale in half-point increments that qualifies disability in participants with MS. It consists of 8 ordinal rating scales assessing seven functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation. EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS).
  units on a scale | 2.67 (1.25) | 2.63 (1.37) | 2.64 (1.18) | 2.65 (1.26)
Dose Level of Interferon-beta (IFN-beta) Based on IVRS [Number; unit: participants]
  High dose | 120 | 128 | 120 | 368
  Low dose | 57 | 50 | 59 | 166

OUTCOME MEASURES:

1. Primary Outcome: Annualized Relapse Rate (ARR) (Poisson Regression Estimates)
Description: ARR is the total number of confirmed relapses that occurred during the treatment period divided by the total number of patient-years treated. Each episode of relapse (appearance, or worsening of a clinical symptom that was stable for at least 30 days, that persisted for a minimum of 24 hours in the absence of fever) was to be confirmed by an increase in Expanded Disability Status Scale (EDSS) score or Functional System scores. To account for the different treatment durations among participants, a Poisson regression model with robust error variance was used (total number of confirmed relapses as response variable; log-transformed treatment duration as "offset" variable; treatment group, region of enrollment and IFN-beta dose stratum, and number of relapses in the year prior to randomization as covariates).
Time Frame: Up to a maximum of 108 weeks depending on time of enrollment
Population: Intent-to-treat (ITT) population: all randomized and treated participants. Participants were considered in the treatment group to which they were randomized regardless of the drug they actually received.
Measure: Number (95% Confidence Interval); unit: relapses per patient-year
Arm/Group | Placebo + IFN-beta | Teriflunomide 7 mg + IFN-beta | Teriflunomide 14 mg + IFN-beta
Number analyzed (Participants) | 175 | 178 | 179
relapses per patient-year | 0.298 [0.206 to 0.432] | 0.242 [0.152 to 0.386] | 0.238 [0.162 to 0.351]

2. Secondary Outcome: Brain Magnetic Resonance Imaging (MRI) Assessment: Number of Gadolinium Enhancing (Gd-enhancing) T1-lesions Per Scan (Poisson Regression Estimates)
Description: Number of Gd-enhancing T1-lesions per scan is the total number of Gd-enhancing T1-lesions that occurred during the treatment period divided by the total number of scans performed during the treatment period. To account for the different number of scans among participants, a Poisson regression model with robust error variance was used (total number of Gd-enhancing T1-lesions as response variable; log-transformed number of scans as offset variable; treatment group, region of enrollment, IFN-beta dose stratum and baseline number of Gd-enhancing T1-lesions as covariates).
Time Frame: Up to a maximum of 108 weeks depending on time of enrollment
Population: ITT population as previously defined but including only participants who had post-baseline data.
Measure: Number (95% Confidence Interval); unit: lesions per scan
Arm/Group | Placebo + IFN-beta | Teriflunomide 7 mg + IFN-beta | Teriflunomide 14 mg + IFN-beta
Number analyzed (Participants) | 151 | 142 | 151
lesions per scan | 0.542 [0.344 to 0.855] | 0.257 [0.127 to 0.523] | 0.158 [0.070 to 0.360]

3. Secondary Outcome: Time to 12-Week Sustained Disability Progression
Description: The 12-week sustained disability progression was defined as an increase from baseline of at least 1-point in EDSS score (at least 0.5-point for participants with baseline EDSS score >5.5) that persisted for at least 12 weeks. Probability of disability progression was to be estimated using Kaplan-Meier method.
Time Frame: Up to a maximum of 108 weeks depending on time of enrollment
Population: Data for this outcome was not analyzed because of insufficient data after early study termination.
Arm/Group | Placebo + IFN-beta | Teriflunomide 7 mg + IFN-beta | Teriflunomide 14 mg + IFN-beta
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Brain MRI Assessment: Volume of Gd-enhancing T1-lesions Per MRI Scan
Description: Total volume of Gd-enhancing T1-lesions per scan is the sum of the volumes of Gd-enhancing T1-lesions observed during the treatment period divided by the total number of scans performed during the treatment period.
Time Frame: Up to a maximum of 108 weeks depending on time of enrollment
Population: ITT population as previously defined but including only participants who had post-baseline data.
Measure: Number; unit: milliliters per scan
Arm/Group | Placebo + IFN-beta | Teriflunomide 7 mg + IFN-beta | Teriflunomide 14 mg + IFN-beta
Number analyzed (Participants) | 151 | 142 | 151
milliliters per scan | 0.045 | 0.009 | 0.01

5. Secondary Outcome: Brain MRI Assessment: Change From Baseline in Total Lesion Volume (Burden of Disease) at Week 24
Description: The total lesion volume (burden of disease) is the total volumes of hyperintense on T2 plus hypointense on T1 as measured by MRI scan. Least-square means were estimated using a Mixed-effect model with repeated measures (MMRM) on cubic root transformed volume data with factors for treatment, region, IFN-beta dose stratum, visit, treatment-by-visit interaction, cubic root transformed baseline burden of disease, and baseline-by-visit interaction.
Time Frame: Baseline, Week 24
Population: ITT population as previously defined but including only participants who had post-baseline data.
Measure: Least Squares Mean (Standard Error); unit: milliliter
Arm/Group | Placebo + IFN-beta | Teriflunomide 7 mg + IFN-beta | Teriflunomide 14 mg + IFN-beta
Number analyzed (Participants) | 142 | 132 | 141
milliliter | -0.008 (0.021) | -0.011 (0.021) | -0.044 (0.020)

6. Secondary Outcome: Time to Relapse: Kaplan-Meier Estimates of the Probability of no Relapse at Week 24, 48, and 72
Description: Probability of no relapse at 24, 48 and 72 weeks was estimated using Kaplan-Meier method on the time to relapse defined as the time from randomization to first EDSS confirmed relapse. Participants free of confirmed relapse (no EDSS confirmed relapse observed on treatment) were censored at the date of the last study drug intake. Kaplan-Meier method consists in computing probabilities of non-occurrence of event at any observed time of event and multiplying successive probabilities for time <=t by any earlier computed probabilities to estimate the probability of being event-free for the amount of time t.
Time Frame: Up to a maximum of 108 weeks depending on time of enrollment
Population: ITT population as previously defined.
Measure: Number (95% Confidence Interval); unit: percent probability of no relapse
Arm/Group | Placebo + IFN-beta | Teriflunomide 7 mg + IFN-beta | Teriflunomide 14 mg + IFN-beta
Number analyzed (Participants) | 175 | 178 | 179
percent probability of no relapse
  Percent probability of no relapse at Week 24 | 81.9 [75.8 to 88.0] | 86.8 [81.4 to 92.1] | 87.1 [81.8 to 92.3]
  Percent probability of no relapse at Week 48 | 67.3 [58.8 to 75.8] | 80.6 [73.3 to 87.8] | 80.8 [73.9 to 87.7]
  Percent probability of no relapse at Week 72 | 58.3 [45.4 to 71.2] | 78.2 [69.8 to 86.6] | 73.1 [62.2 to 83.9]

7. Secondary Outcome: Change From Baseline in Fatigue Impact Scale (FIS) Total Score at Week 24
Description: FIS is a participant-reported scale that qualifies the impact of fatigue on daily life in participants with MS.
Time Frame: Baseline, Week 24
Population: Data for this outcome was not analyzed because of insufficient data after early study termination.
Arm/Group | Placebo + IFN-beta | Teriflunomide 7 mg + IFN-beta | Teriflunomide 14 mg + IFN-beta
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline in Short Form Generic Health Survey - 36 Items, Version 2 (SF-36v2) Summary Scores at Week 24
Description: SF-36 scale is a generic, self-administered, health-related quality-of-life (QOL) instrument.
Time Frame: Baseline, Week 24
Population: Data for this outcome was not analyzed because of insufficient data after early study termination.
Arm/Group | Placebo + IFN-beta | Teriflunomide 7 mg + IFN-beta | Teriflunomide 14 mg + IFN-beta
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Resource Utilization When Relapse
Description: Resource utilization each time a participant experiences an MS relapse, specifically the number of hospitalizations, the number of over night spent in the hospital and number of intensive care admissions if hospitalized were to be reported.
Time Frame: Up to a maximum of 108 weeks depending on time of enrollment
Population: Data for this outcome was not analyzed because of insufficient data after early study termination.
Arm/Group | Placebo + IFN-beta | Teriflunomide 7 mg + IFN-beta | Teriflunomide 14 mg + IFN-beta
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Overview of Adverse Events (AEs)
Description: AEs are any unfavorable and unintended sign, symptom, syndrome, or illness observed by the investigator or reported by the participant during the study.
Time Frame: First study drug intake up to 28 days after last study drug intake, for up to 112 weeks
Population: Safety population: all randomized and treated participants. Participants were included in the treatment group according to the drug actually received.The participant randomized to Teriflunomide 14 mg group who received Teriflunomide 7 mg was analyzed in the Teriflunomide 7 mg group.
Measure: Number; unit: participants
Arm/Group | Placebo + IFN-beta | Teriflunomide 7 mg + IFN-beta | Teriflunomide 14 mg + IFN-beta
Number analyzed (Participants) | 175 | 179 | 178
participants
  Any AE | 119 | 140 | 140
  Any Serious AE | 8 | 13 | 14
  Any AE Leading to Death | 0 | 0 | 0
  Any AE Leading to Study Drug Discontinuation | 9 | 16 | 22

11. Other Pre Specified Outcome: Liver Function: Number of Participants With Potentially Clinically Significant Abnormalities (PCSA)
Description: PCSA values are abnormal values considered medically important by the Sponsor according to predefined criteria based on literature review. Hepatic parameters thresholds were defined as follows: Alanine Aminotransferase (ALT) >3, 5 or 10 Upper Limit of Normal (ULN); Aspartate Aminotransferase (AST) >3, 5 or 10 ULN; Alkaline Phosphatase >1.5 ULN; Total Bilirubin (TB) >1.5 ULN; and ALT >3 ULN and TB >2 ULN.
Time Frame: First study drug intake up to 28 days after last study drug intake, for up to 112 weeks
Population: Safety population as previously defined but including only participants who had post-baseline values.
Measure: Number; unit: participants
Arm/Group | Placebo + IFN-beta | Teriflunomide 7 mg + IFN-beta | Teriflunomide 14 mg + IFN-beta
Number analyzed (Participants) | 174 | 179 | 178
participants
  ALT >3 ULN | 6 | 9 | 9
  ALT >5 ULN | 1 | 6 | 5
  ALT >10 ULN | 1 | 3 | 2
  AST >3 ULN | 3 | 4 | 4
  AST >5 ULN | 2 | 3 | 3
  AST >10 ULN | 1 | 2 | 0
  Alkaline Phosphatase >1.5 ULN | 0 | 2 | 0
  TB >1.5 ULN | 2 | 0 | 2
  ALT >3 ULN and TB >2 ULN | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All AEs were collected regardless of seriousness or relationship to the drug, spanning from signature of the Informed Consent up to the last visit.
Description: The analysis was performed on the safety population and included all AEs that developed or worsened from first study drug intake up to 28 days after last study drug intake, for up to 112 weeks. Participants were included in the treatment group according to the drug actually received.
Arm/Group | Placebo + IFN-beta | Teriflunomide 7 mg + IFN-beta | Teriflunomide 14 mg + IFN-beta
Serious Adverse Events (participants affected / at risk) | 8/175 | 13/179 | 14/178
Other Adverse Events (participants affected / at risk) | 85/175 | 94/179 | 104/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + IFN-beta (N=175) | Teriflunomide 7 mg + IFN-beta (N=179) | Teriflunomide 14 mg + IFN-beta (N=178)
Cystitis (Infections and infestations) | 0 | 0 | 1
Testicular seminoma (pure) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 1 | 2 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + IFN-beta (N=175) | Teriflunomide 7 mg + IFN-beta (N=179) | Teriflunomide 14 mg + IFN-beta (N=178)
Gastroenteritis (Infections and infestations) | 0 | 1 | 9
Nasopharyngitis (Infections and infestations) | 20 | 21 | 20
Upper respiratory tract infection (Infections and infestations) | 12 | 9 | 9
Urinary tract infection (Infections and infestations) | 5 | 10 | 4
Neutropenia (Blood and lymphatic system disorders) | 4 | 8 | 10
Dizziness (Nervous system disorders) | 5 | 8 | 9
Headache (Nervous system disorders) | 14 | 19 | 22
Hypertension (Vascular disorders) | 8 | 7 | 15
Diarrhoea (Gastrointestinal disorders) | 6 | 16 | 20
Nausea (Gastrointestinal disorders) | 9 | 18 | 12
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 11 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 8 | 7
Influenza like illness (General disorders) | 8 | 9 | 4
Alanine aminotransferase increased (Investigations) | 15 | 16 | 26

LIMITATIONS AND CAVEATS:
The early termination of study with reduced sample size and participant follow-up impacts the power and interpretability, and limits the ability to assess the overall benefit/risk of adjunctive therapy. Termination was not due to any safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.